CLINICAL TRIAL: NCT02509871
Title: Study of Body Composition in Patients Treated by Adjuvant Hormonal Therapy for Breast Cancer
Brief Title: Study of Body Composition in Patients Treated by Adjuvant Hormonal Therapy for Breast Cancer (MetaCa2)
Acronym: MetaCa2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A00633-46
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Hormonal Therapy; Breast Cancer
Keywords: Body composition
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body composition measurement (Other): DXA, impedance
  Interventions: Other: Body composition measurement

INTERVENTIONS:
Other: Body composition measurement — DXA, impedance

SUMMARY:
This cross-sectional study of pathophysiology will bring additional informations on body composition of patients treated by adjuvant hormonal therapy for breast cancer. This is a complementary study of Metaca study (AU882).

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* patients requiring hormonal treatment
* WHO performance status 0-2
* patients initially included in MetaCa (AU882) protocol
* Affiliation to a social security scheme (or be the beneficiary of such a plan)
* patients who signed the informed consent form

Exclusion Criteria:

* patients witg relapse, with metastases or other cancer
* concurrent treatment with a drug test, or participation in a clinical trial within < 30 days
* patients carrying an electronic medical device (eg pacemaker)
* patients who refused to sign the consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measure of body composition | After more than a year of hormonal therapy
  To obtain additional data to those of Metaca study (AU882) to assess changes in body composition (fat mass, lean body mass in Kg) in women with breast cancer and treated with adjuvant hormonal therapy following chemotherapy

SECONDARY OUTCOMES:
Evaluation of the distribution of abdominal fat by measuring the waist and hip circumference | After more than a year of hormonal therapy
Assessment of anxiety and depression scores measured by Questionnaire HAD | After more than a year of hormonal therapy
  Questionnaire HAD
Evaluation of quality of life measured by Questionnaire (QLQ-C30) | After more than a year of hormonal therapy
  Questionnaire (QLQ-C30)
Evaluation of the time sitting measured by Questionnaire IPAQ | After more than a year of hormonal therapy
  Questionnaire IPAQ
Evaluate the change in body composition longitudinally from the data of the study Metaca | Between after 1 and 6 months after chemotherapy and after more than a year of hormonal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, MD, PhD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France

REFERENCES:
- [Result] Ginzac A, Thivat E, Mouret-Reynier MA, Dubray-Longeras P, Van Praagh I, Passildas J, Abrial C, Kwiatkowski F, Boirie Y, Duclos M, Morio B, Gadea E, Durando X. Weight Evolution During Endocrine Therapy for Breast Cancer in Postmenopausal Patients: Effect of Initial Fat Mass Percentage and Previous Adjuvant Treatments. Clin Breast Cancer. 2018 Oct;18(5):e1093-e1102. doi: 10.1016/j.clbc.2018.06.010. Epub 2018 Jun 18. PMID 30417829